CLINICAL TRIAL: NCT04495686
Title: An Innovative Supportive Care Model for Dementia and Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carol Manning, Harrison Distinguished Teaching Professor of Neurology, Vice Chair for Faculty Development, Director Memory Disorders Clinic, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-HSR #15372
Record Dates: First submitted 2020-05-18; First posted 2020-08-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Dementia, Mixed; Dementia Mild; Dementia Moderate; Traumatic Brain Injury; Alzheimer Disease
Keywords: dementia; traumatic brain injury; caregiver; alzheimers
MeSH Terms: conditions — Mixed Dementias; Brain Injuries, Traumatic; Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Caregiver PWD-ADRD TCCI (Experimental): Participants in the Caregiver PWD-ADRD telehealth care coordination intervention (TCCI) group will complete a 12-month telehealth-delivered care coordination program with an assigned dementia care coordinator.
  Interventions: Behavioral: Telehealth-delivered Care Coordination Program
- Caregiver for PWD-ADRD (BMT) (No Intervention): Participants in the Caregiver PWD-ADRD best medical treatment (BMT) group will not receive care coordination.
- Caregiver for PWD-TBI TCCI (Experimental): Participants in the Caregiver PWD-TBI telehealth care coordination intervention (TCCI) group will complete a 12-month telehealth-delivered care coordination program with an assigned dementia care coordinator.
  Interventions: Behavioral: Telehealth-delivered Care Coordination Program
- Caregiver for PWD-TBI (BMT) (No Intervention): Participants in the Caregiver PWD-TBI best medical treatment (BMT) group will not receive care coordination.

INTERVENTIONS:
Behavioral: Telehealth-delivered Care Coordination Program — Participants in the interventional arms of this program will be assigned a Dementia Care Manager (DCM) who will work with caregivers to develop goals and plans that are aimed at providing the best support possible, specific to your needs. These services include supportive counseling, education on dementia, information and referrals to community-based organizations, behavioral symptom management training and assistance with finding available community and government-sponsored programs.
  DCM's will meet with you at least once monthly and will be available if you need assistance between meetings. At the first meeting, your DCM will explain the questionnaires you will take and how to use the technology in the program. They will then provide a link, via email, where you will download the free teleconferencing software that will be used throughout the program. Questionnaires will then be sent via email invitations through a secure survey platform.
  Arms: Caregiver PWD-ADRD TCCI; Caregiver for PWD-TBI TCCI

SUMMARY:
There are an increasing number of people in the U.S. with Alzheimer's disease and other dementias. Traumatic brain injuries (TBIs) are also common among both civilians and military personnel, and TBIs increase a person's risk for dementia. Providing care for a person with dementia is stressful. Dementia caregivers can experience difficulties including stress, depression, and reduced quality of life. Coordinated dementia care is known to benefit people with dementia and their caregivers. However, many caregivers do not have access to these supportive programs.

Our project studies the benefits of telehealth as a new way for caregivers to receive coordinated dementia care services. We will offer 75 caregivers a 12-month caregiver support program delivered using telehealth (for example phones, tablets, computers). Caregivers of both Alzheimer's disease and TBI-related dementia will be included, and the program will be evaluated for effectiveness in both groups as well as in a control group. The information from our study will help improve quality of life for caregivers and individuals with dementia, including military members and Veterans. Our results will also help both civilian and military health professionals develop effective programs to support families living with dementia. Policy makers and organizational leaders can use the information to fund programs that best help families and communities facing dementia and TBI dementia.

DETAILED DESCRIPTION:
More than 150,000 Virginians live with dementia. Most persons with dementia (PWD) are cared for by an unpaid family caregiver. These caregivers' provision of daily assistance to PWD is a critical part of the state's dementia care capabilities. Caregivers of PWD experience an array of negative biopsychosocial impacts related to their caregiving responsibilities that undermine their own well-being and their care capacity. They are often unprepared to manage the behavioral symptoms of dementia (BSD); unmanaged symptoms are associated with increased use of emergency care and institutional placement, which are burdensome outcomes for PWD, families, and public health systems.

An emergent body of research associates traumatic brain injury (TBI) with increased dementia risk. Veterans with a history of TBI are therefore at increased risk of developing dementia, putting their family members at risk for the established negative impacts of caregiving. Coordinated care programs have proven beneficial for both members of the dementia caregiving dyad, yet access barriers remain. Many caregivers have competing role responsibilities that conflict with consistent dementia care access, others are located in rural areas without access to specialized dementia care.

To surmount access barriers and countervail the negative impacts of caregiving, we propose an innovative, non-pharmacological intervention: a telehealth-delivered dementia care coordination program that provides family and caregiver support and will improve the quality of life (QoL) for both caregivers and PWD. A goal of our project is to fill an existing service gap by providing coordinated dementia care to an underserved population: caregivers of persons with TBI dementia.

Our study will test three primary hypotheses: 1) Caregivers of persons with dementia who participate in the telehealth care coordination program will experience greater improvements in study caregiver outcomes (depression, burden, reactions to BSD and QoL) than caregivers of PWD receiving best medical treatment (BMT); 2) Caregivers who participate in the program will experience greater satisfaction with care than caregivers in the BMT group; 3) The program will comparable benefits for caregivers of persons with Alzheimer's disease and related dementia (PWD-ADRD) and persons with TBI dementia (PWD-TBI).

In addition, our study includes three exploratory hypotheses: 1) Certain caregiver characteristics (external locus of control; lower self-efficacy, sense of hope, and self-perceived caregiver aptitude) will be negatively associated with improvements in caregiver study outcomes; 2) Caregivers in the intervention group will experience greater reductions in emergency/unnecessary health care utilization then caregivers in the BMT group; 3) The intervention will impart sustained caregiver benefits in primary study outcomes.

Project specific aims include: 1) Evaluate the benefits of a telehealth-delivered care coordination program intervention for caregivers of PWD relative to best medical treatment; 2) Evaluate the impact of the intervention on caregiver satisfaction; 3) Determine the comparative effectiveness of the care coordination program between caregivers of persons with ADRD those with TBI dementia; 4) Explore caregiver characteristics that influence intervention outcomes (burden, depression, QoL, responses to BSD); and 5) Investigate whether the intervention reduces emergency and unplanned health care utilization.

Our research strategy is a prospective, randomized, unblinded study investigating the benefits of a 12-month telehealth-delivered dementia care coordination intervention, with follow up assessments to examine the longevity of the intervention impacts. We will enroll 3 study groups: 50 caregivers of PWD-ADRD receiving the telehealth coordinated care intervention; 50 caregivers of PWD-ADRD receiving best medical treatment, and 25 caregivers of PWD-TBI receiving the intervention. We will collect baseline,12-, and 18-month data to examine intervention effectiveness on caregiver study outcomes and test the prolonged intervention effects.

Our study uses an innovative telehealth approach to provide care for families living with dementia. Family support has important implications at the individual, family, community, and national level. Strategies to reduce caregiver burden and improve QoL for civilian and military families can lead to greater satisfaction with care and prolong caregivers' capacity to keep their loved ones at home, reducing burdens on public payment systems, including the VA. Dissemination of study results will inform state and local policy and finance decisions that can help improve the lives of the growing population of persons with dementia or TBI dementia.

ELIGIBILITY:
Caregiver Inclusion Criteria:

* Must be at least 18 years of age
* Self-identified primary caregiver for a community-dwelling patient with dementia (PWD)
* Must be an unpaid caregiver
* Basic spoken and written English language skills

Caregiver Exclusion Criteria:

* Unwilling or unable to fulfill the requirements of the study
* Any condition which would make the caregiver, in the opinion of the investigator, unsuitable for the study
* No access to high-speed/broadband internet service capable of operating study teleconferencing software available

Patient with Dementia Inclusion Criteria:

* aged 55 years or older
* Diagnosis of mild cognitive impairment (MCI) or Alzheimer's disease and related dementias (ADRD)
* Mild to moderate dementia, including mixed dementia
* 0-1 appointments in the multi-disciplinary long-term University of Virginia (UVA) Memory Disorder follow-up clinic (MDC)

Patient with Dementia and TBI Inclusion Criteria:

* aged 21 years or older
* Diagnosis of major neurocognitive disorder (MND), mild neurocognitive disorder, or Alzheimer's disease and related dementias (ADRD)
* Diagnosis of mild to moderate dementia, including mixed dementia
* Diagnosed with mild complicated, moderate or sever traumatic brain injury (TBI)
* TBI event at or after the age of brain maturity, ≥25 years of age

No exclusion criteria for patients with dementia and/or traumatic brain injury.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Depression: Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) | Change outcome measure at Baseline and 12 months and 18 months
  The CESD-R assesses self-reported symptoms of depression. The revised version was developed to reflect current understanding of psychiatric depressive symptoms. The revised 20-item version is highly correlated with the original CESD, demonstrating test validity.
Caregiver Burden: Zarit Burden Interview (ZBI) | Change outcome measure at Baseline and 12 months and 18 months
  The ZBI is a 22-item caregiver self-report measure assessing degree of caregiver burden in caregivers of PWD. The validated ZBI questions include measures of caregivers' health, finances, social supports, and psychological well-being.
Caregiver Reactions to the Behavioral Symptoms of Dementia: Revised Memory and Behavior Problem Checklist (RMBPC) | Change outcome measure at Baseline and 12 months and 18 months
  The RMBPC is a 24-item, caregiver-reported measure that assesses the frequency of problematic behaviors in patients with dementia and the severity of caregivers' reactions to these behaviors. The reliability and validity of the RMBPC have been established.
Quality of Life: WHO (Five) Well-Being Index (WHO-5) | Change outcome measure at Baseline and 12 months and 18 months
  The WHO-5 contains five questions that measure well-being; scores range from 0-25, with higher scores representing higher QoL. The WHO-5 is a validated tool that has been used successfully as an outcome measure in clinical trials across a wide range of study fields.
Satisfaction with Care: Caregiver Satisfaction Survey (CSS) | Change outcome measure at 12 months and 18 months
  The CSS is an investigator-developed survey that assesses satisfaction with care services.

SECONDARY OUTCOMES:
Healthcare Resource Utilization: Resource Utilization in Dementia, (RUD) questionnaire version 4.0. | Baseline, 12 months
  The RUD v4.0 is a standardized, widely used instrument to collect resource use data in dementia. Caregivers are asked to report resource utilization for both themselves and the person for whom they are caring.
Neuropsychiatric Symptoms and Caregiver Reactions: Neuropsychiatric Inventory Questionnaire (NPI-Q). | Baseline, 12 months
  NPI is a validated instrument measuring 12 subdomains of psychopathology (e.g. delusions, agitation/aggression, nighttime behavior) for persons with dementia as assessed by their caregivers. Content and concurrent validity as well as inter-rater and test-retest reliability have been established.
Anxiety: Geriatric Anxiety Inventory (GAI). | Baseline, 12 months
  The GAI comprises 20 items that measure self-reported symptoms of anxiety in older adults. The GAI has established internal consistency, test-retest reliability, validity, and sensitivity.
Dementia Knowledge: Dementia Knowledge Assessment Tool Version 2 (DKAT2). | Baseline, 12 months
  The DKAT2 assesses family caregivers' foundational-level knowledge of dementia and covers 2 domains: dementia and its progress, and dementia support and care. The DKAT2's internal consistency, reliability, and content validity have been established.
Preparedness for Caregiving: Preparedness for Caregiving Scale (PCS). | Baseline, 12 months
  The PCS is an 8-item self-report instrument that gauges how well caregivers believe they are prepared for multiple domains of caregiving, including providing physical care and emotional support, setting up home-based support services, and handing caregiver stress. The scale's validity and reliability are established.
Self-Efficacy: General Self-Efficacy scale (GSE). | Baseline, 12 months
  The GSE is a validated, reliable self-report measure of self-efficacy. Scores on the 10-item scale range from 10-40, with higher scores indicating higher self-efficacy.
Optimism/Pessimism: Life-Orientation Test-Revised (LOT-R) | Baseline, 12 months
  The LOT-R is a 10-item test that quantifies optimism. The test has predictive and discriminate validity and can distinguish optimism from constructs such as depression, self-esteem, and self-mastery.
Basic Activities of Daily Living: Katz Index of Independence in Activities of Daily Living (Katz). | Baseline, 12 months
  The KATZ is a validated measure of function used to objectively evaluate chronically ill and aging populations. The measure ranks overall performances in six functions that indicate independence in 6 basic activities of daily living: bathing, dressing, toileting, transferring, feeding, and continence.
Instrumental Activities of Daily Living: Lawton Instrumental Activities of Daily Living Scale (Lawton). | Baseline, 12 months
  The Lawton scale measures a person's level of independence in the completion of instrumental activities of daily living. The validated scale detects functional decline across 8 domains: shopping, food preparation, taking medications, ability to handle finances or use a telephone, laundry, housekeeping, and transportation.
Quality of Life in PWD: Quality of Life in Alzheimer's Disease (QoL-AD). | Baseline, 12 months
  The QoL-AD assesses quality of life reported by older adults with cognitive impairment and their caregivers. The validated 10-minute test has good internal and test-retest reliability. The 13 items were developed based on Lawton's scale for QoL domains and feedback from individuals with dementia and their caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Manning, Ph.D., Principal Investigator — University of Virginia Department of Neurology
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include self-reported demographic information and behavioral data from well-validated questionnaires. Because subjects will be recruited within the University of Virginia Memory and Aging Care Clinic and provided clinical services through this clinic that intersect with their participation in this study, we will be collecting identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. We are specifically concerned about the potential for negative consequences subsequent to deductive disclosure due to the sensitive nature of the behavioral and diagnostic information being obtained in this study and the potential for these consequences to affect both the study subject and the PWD for whom they provide care.
Supporting Information: SAP, CSR
Time Frame: We will make this final research data available by the time of publication of the main findings from the final dataset.
Access Criteria: we will make the final research data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Gallagher VT, Reilly SE, Arp A, Rossetti A, Thompson R, Manning CA. Randomized clinical trial of the individualized coordination and empowerment for care partners of persons with dementia (ICECaP) intervention: impact on preparedness for caregiving. Aging Clin Exp Res. 2025 Mar 1;37(1):64. doi: 10.1007/s40520-025-02959-z. PMID 40021531
- [Derived] Thompson RC, Gallagher VT, Reilly SE, Arp AM, Manning CA. Individualized Coordination and Empowerment for Care Partners of Persons with Dementia (ICECaP): Feasibility and acceptability. Contemp Clin Trials. 2025 Jan;148:107770. doi: 10.1016/j.cct.2024.107770. Epub 2024 Dec 2. PMID 39631536
- [Derived] Gallagher VT, Arp A, Thompson R, Rossetti A, Patrie J, Reilly SE, Manning CA. Randomized Clinical Trial of ICECaP (Individualized Coordination and Empowerment for Care Partners of Persons with Dementia): Primary Mental Health and Burden Outcomes. medRxiv [Preprint]. 2024 Aug 16:2024.08.15.24312041. doi: 10.1101/2024.08.15.24312041. PMID 39185526